CLINICAL TRIAL: NCT06069453
Title: Intravesical Hyaluronic Acid Sodium Salt and Hydeal-D for Relief of Storage Lower Urinary Tract Symptoms (LUTS) After Trans-urethral Resection of Bladder Tumor (TURBT) for Non-muscle Invasive Bladder Cancer (NMIBC). Monocentric, Randomized, Controlled Investigation.
Brief Title: Hyaluronic Acid Sodium Salt and Hydeal-D in the Management of LUTS After TURBT for NMIBC.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UQP6-19-01
Record Dates: First submitted 2023-09-08; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, controlled investigation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Solution containing Hyaluronic Acid (HA) sodium salt and Hydeal-D
  Interventions: Device: Hyaluronic Acid (HA) sodium salt and Hydeal-D
- Group B (No Intervention): standard management according to institutional protocol

INTERVENTIONS:
Device: Hyaluronic Acid (HA) sodium salt and Hydeal-D — intravesical solution containing Hyaluronic Acid (HA) sodium salt and Hydeal-D
  Arms: Group A

SUMMARY:
This will be an open-label, prospective, single-centre, randomised, controlled, parallel-group medical device investigation. The investigational plan will include four visits in total at the investigational site. One visit (Visit 2) will consist in the hospitalisation period and will last 3/4 days. Patients will be admitted to hospital in the day preceding the TURBT (Day -1; in case the TURBT is programmed in the morning) or in the day of the TURBT (Day 0; in case the TURBT is programmed in the afternoon) and will stay in the hospital for 3/4 days after the intervention (performed on Day 0). Patients will then be discharged, if considered as appropriate based on Investigator's judgment, following the removal of the catheter and the first clear urination. Patients will be asked to remain in the same geographic area of the investigational site up to the end of study visit.

DETAILED DESCRIPTION:
The following visits/activities will be performed:

* Visit 1: the screening visit will be performed between 60 and 14 days before the TURBT (Day -60/-14);
* Visit 2 (hospitalisation): patients will be admitted to hospital in the day preceding the TURBT or in the day of the TURBT and will be randomised to the assigned treatment group. TURBT will be performed on Day 0. The first treatment with the investigational device will be performed within 6 hours from the end of TURBT. The catheter will be removed at Day 2 ± 1 if considered as appropriate based on Investigator's judgment, following the first clear urination). The second treatment with the investigational device will be performed just before the removal of the catheter and the discharge from hospital.
* Visit 3: a follow-up visit will be performed at Day 5 ± 1 (i.e. 3 days after catheter removal);
* Visit 4: the end of study visit will be performed at Day 25 ± 4.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females patients aged ≥ 18 years old;
2. Patients with suspected clinical diagnosis of primary or secondary single or multiple, any size, NMIBC scheduled for TURBT;
3. Female patients with child-bearing potential must not be pregnant or lactating, and willing to use adequate contraception for the duration of study. Note: to be considered females of non-child-bearing potential, females must be surgically sterile or postmenopausal as documented in medical history for at least 1 year.

   Highly effective birth control methods include: combined hormonal contraception (containing estrogens and progestogen) associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence.
4. Patients available to remain in the same geographical area of the investigational site from the hospitalisation to the end of the investigation;
5. Patients able to understand and comply with the requirements of the study and voluntarily provide written informed consent.

Exclusion Criteria:

1. Patients with Schistosoma haematobium infestation or neurologenic bladder;
2. Patients having received (in the three months before the screening) previous treatment with neurotoxic drugs (e.g. vanilloids, ovanil, botulinum toxin, etc.) or pelvic irradiation, which could interfere with sensory functions;
3. Patients with indication for early instillation due to new treatment guideline;
4. Patients with any potential interfering factors for LUTS evaluation, such as obstruction, nocturnal polyuria strictures, neurogenic bladder, detrusor over/under capacity;
5. Patients with clinically relevant comorbidities that could potentially interfere with study evaluations, such as diabetes, renal disease and cardiac failure;
6. Patients with presence of other serious gastrointestinal, renal, hepatic, pulmonary, cardiovascular or neurological disease that could adversely affect the safety of the study treatment or the patient's ability to comply with investigation requirements;
7. Patients on treatment or having received (in 30 days before screening) the following anticholinergic drugs: oxybutinin, tolterodine, fesoterodine, darifenacin, trospium and beta-3 adrenoreceptor agonist;
8. Patients with known or suspected allergy, hypersensitivity or intolerance to hyaluronic acid and/or any other component of the investigational device;
9. Patients with hypersensitivity to local anaesthetics or other drugs used for the procedure;
10. Women who are pregnant or breastfeeding or women who could become pregnant and are not using effective contraception;
11. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the investigation;
12. Patients who have used any investigational drug or device in an investigational protocol in the past 3 months;
13. Patients who have been previously enrolled in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of severity rate of storage symptoms (frequency, urgency, nocturia) compared to control group | 3 days after catheter removal
  Severity of storage symptoms will be evaluated through a patient's bladder diary

SECONDARY OUTCOMES:
Evaluation of severity rate of storage symptoms (frequency, urgency, nocturia) compared to control group | 25 days
  Severity of storage symptoms will be evaluated through patient's bladder diary
Evaluation of changes from baseline in severity of urinary symptoms compared to control group | 25 days
  Change from baseline (Day -1) in severity of urinary symptoms will be evaluated by IPSS. Scores obtained in the group of patients treated with Hydeal Cyst® will be compared with scores obtained in the control group. Storage and voiding symptoms will be also estimated in both arms by IPSS-s and IPSS-v subscores.The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic) and the overall intensity of urinary symptoms is categorised in mild (score 1-7), moderate (score 8-19) and severe (score 20-35).
Evaluation of changes from baseline in severity rate of urinary symptoms compared to control group | 25 days
  Change from baseline in severity and frequency of urinary symptoms, as evaluated by ICIQ-MLUTS in males and ICIQ-FLUTS in females. Scores obtained in the group of patients treated with Hydeal Cyst® will be compared with scores obtained in the control group.The ICIQ is a questionnaire for evaluating male lower urinary tract symptoms and impact on quality of life (QoL) .All items are evaluated using a score rated 0-4 for frequency and a score 0-10 for bothering, with higher scores corresponding to higher severity of symptoms.
Evaluation of changes from baseline in severity of pelvic pain compared to control group | 25 days
  Change from baseline in severity of pelvic pain, as evaluated by means of a 0-100 mm visual analogue scale (VAS). Scores in the group of patients treated with Hydeal Cyst® will be compared with scores obtained in the control group.
Duration of catheter implant as time of permanence of cathether implanted compared to control group | 49 hours
  The time (hours) of permanence of catheter implanted will be counted for every patient and will be codified in classes (< 47 hours, 48 ± 1 hours, > 49 hours). The frequencies in the group of patients treated with Hydeal Cyst® will be calculated and compared with those of the control group. The analysis of the duration of catheter implant will be performed by means of a Chi-square test or a Fisher's Exact test on the analysis of classes (< 47 hours, 48 ± 1 hours, > 49 hours).
Rescue medication consumption after surgery compared to control group | 25 days
  The proportion of users and the amount of used rescue medication in the treated-group of patients with Hydeal Cyst® will be compared with those of the control group.
Evaluation of quality of life using the EuroQoL-5D compared to control group | 25 days
  Quality of life will be evaluated using the EQ-5D-5L (QoL), as mean scores of patients treated with Hydeal Cyst® compared with scores of control group.The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Number of participants with treatment-related adverse events compared to the control group | 25 days
  Adverse Events (AEs) encountered will be reported and documented in the AE page of the e-CRF, whether considered to be related to the investigational device or not. If the Adverse Event is serious, the Serious Adverse Event Form must also be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Giordan, Study Director — Fidia Farmaceutici s.p.a.
Locations (1):
- Humanitas Research Hospital, Rozzano, Mi, Italy

IPD SHARING:
Plan to Share IPD: No